CLINICAL TRIAL: NCT04753112
Title: Treatment of Pulmonary Hypertension With Angiotensin II Receptor Blocker and Neprilysin Inhibitor in Patients With Heart Failure With Preserved Ejection Fraction Monitored With the CardioMEMS Device (ARNIMEMS-HFpEF)
Brief Title: Treatment of PH With Angiotensin II Receptor Blocker and Neprilysin Inhibitor in HFpEF Patients With CardioMEMS Device
Acronym: ARNIMEMS-HFpEF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICOR-2020-03-PA-ARNIMEMS
Record Dates: First submitted 2021-02-01; First posted 2021-02-15 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; preserved ejection fraction; heart failure
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure | interventions — sacubitril; Valsartan; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Intervention Model Description: 14 participants (the sample size was calculated accepting an alpha risk of 0.05 and a beta risk of 0.2 in a two-sided contrast, to detect a mean PAP difference equal or greater than 4mmHg, assuming a standard deviation of 5mmHg and a 10% loss to follow-up)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): All the subjects will receive sacubitril/valsartan from weeks 6 to 12. From weeks 1-6 and 12-18 patients will be treated with standard therapy for HFpEF according to PA pressures (diuretics and systemic vasodilators if concomitant hypertension).
  All the subjects will also receive longitudinal pulmonary artery pressure monitoring using a previously placed implantable hemodynamic monitor (CardioMEMS device).
  Device: Patients eligible for this study are those with an already implanted CardioMEMS device.
  Drug: Sacubitril/Valsartan Target dose:97/103mg bid
  Interventions: Drug: Sacubitril / Valsartan Oral Tablet [Entresto]

INTERVENTIONS:
Drug: Sacubitril / Valsartan Oral Tablet [Entresto] — Treatment of Pulmonary Hypertension With Angiotensin II Receptor Blocker and Neprilysin Inhibitor

SUMMARY:
This study will assess the impact of sacubitril/valsartan on elevated pulmonary artery (PA) pressures in patients with heart failure (HF) with preserved ejection fraction (HFpEF), measured using a previously implanted hemodynamic monitoring device (CardioMEMS).

DETAILED DESCRIPTION:
Fluid overload leading to increased PA pressure is one of the primary causes of HF related hospitalizations in HFpEF. Signs and symptoms of fluid overload are not sensitive enough to reflect early pathophysiologic changes that increase the risk of decompensation. Elevations in PA pressure may increase several days or weeks before signs and symptoms manifest.

The CardioMEMS device is a small wireless sensor that is permanently implanted in the PA via a catheter inserted through the femoral vein. The sensor measures PA pressure and is paired with a portable electronic transmitter. The system allows patients to wirelessly transmit pressure readings to a secure online database from which treating physicians can access the data and adjust medication in response to PA pressure changes.

The CHAMPION trial was a single blind randomized clinical trial that showed a significant and large reduction in hospitalizations in patients with NYHA class III HF who were managed with a the CardioMEMS device.

More recently, real life clinical practice has confirmed the value of PA pressure-guided therapy for HF. PA pressures were reduced, lower rates of HF hospitalizations and all-cause hospitalization, and low rates of adverse events across a broad range of patients with symptomatic HF and prior HF hospitalizations were reported.

The angiotensin receptor-neprilysin inhibitor (ARNI) led to a reduced risk of hospitalization for HF or death from cardiovascular causes among patients with HF and reduced ejection fraction in the PARADIGM-HF trial. However it did not result in a significantly lower rate of total hospitalizations for HF and death from cardiovascular causes among patients with HF and an ejection fraction of 45% or higher in the PARAGON-HF trial, despite there was suggestion of heterogeneity with possible benefit with sacubitril-valsartan in patients with lower ejection fraction and in women.

ARNI reduced pulmonary pressures and vascular remodeling in an animal model of pulmonary hypertension (PH) and may be appropriate for treatment of PH and right ventricle dysfunction. Data are lacking on the hemodynamic effects of ARNI on pulmonary hypertension in patients with HFpEF.

This study will assess the impact of sacubitril/valsartan on PA pressures measured using an implanted PA monitoring device. The device will be used according to approved indications.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to provide written informed consent.
* Patients ≥18 years of age, male or female, in NYHA Class II- III HFpEF with LVEF > 45% (measured within the past year), and who have no previous LVEF<45%.
* NT-proBNP >200 pg/ml if HF hospitalization in the previous 9 months and> 300 pg/ml if there was no previous HF hospitalization; Three times the values were required in patients with atrial fibrillation.
* CardioMEMS HF System implanted and patient transmitting information regularly and system functioning appropriately.
* Average PAPm >20mm Hg during the 7 days prior to enrollment, including at least 5 daily measurements.
* Systolic BP > 100 mm Hg at most recent clinical assessment.
* Stable, ambulatory patients without the need for change in diuretics and other HF drugs during last week.

Exclusion Criteria:

* eGFR < 30 ml/min/1.73 m2 as measured by CKD-EPI.
* Sacubitril/Valsartan treatment within the past 30 days.
* History of hypersensitivity, intolerance or angioedema to previous renin-angiotensin system (RAS) blocker, ACE inhibitor, ARB, or Entresto.
* Serum potassium > 5.4 mmol/L.
* Acute coronary syndrome, stroke, transient ischemic attack, cardiovascular surgery, PCI, or carotid angioplasty within the preceding 3 months.
* Coronary or carotid artery disease likely to require surgical or percutaneous intervention within 3 months after trial entry.
* Non-cardiac condition(s) as the primary cause of dyspnea.
* Documented untreated ventricular arrhythmia with syncopal episodes within the prior 3 months.
* Symptomatic bradycardia or second or third degree heart block without a pacemaker.
* Hepatic dysfunction, as evidenced by total bilirubin > 3 mg/dl.
* Pregnancy.
* Women who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Change in mPAP With Sacubitril/Valsartan compared to Standard therapy | Time Frame: 0-18 weeks
  Change in Mean Pulmonary Artery Pressure With Sacubitril/Valsartan compared to Standard therapy.

SECONDARY OUTCOMES:
Mean Change in mPAP | 7 days
  Mean Change in mPAP on Sacubitril/Valsartan (7 days after first dose of sacubitril/valsartan).
Change in Distance Walked | Baseline, 6 weeks, 12 weeks, 18 weeks
  Change in Distance Walked During a Standard 6 Minute Walk
Change in NT-proBNP concentration | 6-12-18 weeks
  Change in NT-proBNP (pg/ml)
Change in CA-125 concentration | 6-12-18 weeks
  Change in CA-125 (u/ml)
Change in Soluble ST2 concentration | 6-12-18 weeks
  Change in Soluble ST2 (ng/ml)
Change in the European Quality of Life-5 Dimensions scale | Baseline, 18 weeks
  Minimum value of 5, maximum value of 15. Higher scores mean a worse quality of life.
Change in the short version of the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | Baseline, 18 weeks
  Minimum value of 0, maximum value of 100. Higher scores mean a better quality of life.
Change in Daily Diuretic Dose | Baseline-6-12-18 weeks
  Mean Change in Total Daily Diuretic Dose
Change in E/e' | 6 weeks, 12 weeks, 18 weeks
  Mean Change in diastolic dysfunction echocardiography parameter E/e'
Change in septal e' velocity | 6 weeks, 12 weeks, 18 weeks
  Mean Change in diastolic dysfunction echocardiography parameter Septal e' velocity (m/s)
Change in lateral e' velocity | 6 weeks, 12 weeks, 18 weeks
  Mean Change in diastolic dysfunction echocardiography parameter lateral e' velocity (m/s)
Change in diastolic dysfunction echocardiography parameter tricuspid regurgitation velocity | 6 weeks, 12 weeks, 18 weeks
  Mean Change in diastolic dysfunction echocardiography parameter tricuspid regurgitation velocity (m/s)
Change in diastolic dysfunction echocardiography parameter left atrium volumen index | 6 weeks, 12 weeks, 18 weeks
  Mean Change in diastolic dysfunction echocardiography parameter left atrium volumen index (ml/m2)
Change in the number of B-lines in lung ultrasound LUS | 6 weeks, 12 weeks, 18 weeks
  Mean Change in the number of B-lines in lung ultrasound
Decline in renal function | Baseline-18 weeks
  Decline in renal function (decrease in the estimated glomerular filtration rate of ≥50%, development of end-stage renal disease, or death due to renal failure)
Prespecified adverse events of interest | Baseline-18 weeks
  Hypotension with systolic blood pressure <100 mmHg, hyperkalemia (>5.5mmol/L), and angioedema are prespecified adverse events of interest

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias i Pujol University Hospital, Badalona, Barcelona, Spain